CLINICAL TRIAL: NCT00255541
Title: A 52-Week Randomized, Double-Blind, Parallel-Group, Multi-Centre, Active-Controlled (Glibenclamide) Study to Evaluate the Efficacy, Safety and Tolerability of Tesaglitazar Therapy When Administered to Patients With Type 2 Diabetes
Brief Title: GALLANT 4 Tesaglitazar vs. Glibenclamide
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00028
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Glyburide

INTERVENTIONS:
Drug: Tesaglitazar
Drug: Glibenclamide

SUMMARY:
This is a 52-week randomized, double-blind, parallel-group, multi-center, active-controlled (glibenclamide) study of tesaglitazar in patients with type 2 diabetes, not adequately controlled on diet and lifestyle advice alone during the run-in period. The study comprises a 6 week placebo single blind run in period followed by a 52-week double blind treatment period and a 3-week follow-up period. Tesaglitazar and glibenclamide will be titrated to optimal effect or highest tolerable dose during the first 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580
Dates: Start 2004-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in glycosylated hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
The change in fasting plasma glucose (FPG), insulin, proinsulin and C-peptide
Insulin sensitivity by assessment of change in the calculated variable homeostasis assessment model
Lipid parameters (triglyceride [TG], total cholesterol, high-density lipoprotein cholesterol [HDL C], non-HDL C, low-density lipoprotein cholesterol [LDL C], apolipoproteins [Apo] A-I, Apo B, Apo CIII, free fatty acids, lipoprotein particle size and c
C-reactive protein, LDL C/HDL C ratio and Apo B/Apo A-I ratio
FPG, homeostasis assessment model, insulin, proinsulin, C-peptide
Tumor necrosis factor-alpha, intracellular adhesion molecule-1
Fibrinogen
Urinary albumin excretion
Waist/hip ratio
Responder analyses for HbA1c, FPG, TG, HDL C, total cholesterol, non HDL C and LDL C according to pre-specified values
Proportion of patients reaching pre-specified target levels for HbA1c, FPG, TG, HDL C, non-HDL C and LDL C
Pharmacokinetics of tesaglitazar
Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (66):
- Belgium (7):
  - Research Site, Antwerp
  - Research Site, Braine-l'Alleud
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Merksem
  - Research Site, Sint-Gillis-Waas
  - Research Site, Steenokkerzeel
- Research Site, Shatin, N.T., Hong Kong
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Székesfehérvár
- Italy (14):
  - Research Site, Arenzano
  - Research Site, Chiavari (GE)
  - Research Site, Chieri
  - Research Site, Gubbio (PG)
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Piacenza
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Rho
  - Research Site, Roma
  - Research Site, Udine
- Malaysia (2):
  - Research Site, Kubang Kerian, Kota Bharu
  - Research Site, Kuala Lampur
- Mexico (4):
  - Research Site, México, D.F.
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Veracruz
- Norway (8):
  - Research Site, Ås
  - Research Site, Bergen
  - Research Site, Kongsvinger
  - Research Site, Lysaker
  - Research Site, Oslo
  - Research Site, Skedsmokorset
  - Research Site, Sørumstand
  - Research Site, Trondheim
- Philippines (2):
  - Research Site, Manila
  - Research Site, Pasig
- Poland (7):
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, P³ock
  - Research Site, Toruñ
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, £ód?
- Slovakia (9):
  - Research Site, Bratislava
  - Research Site, Ilava
  - Research Site, Košice
  - Research Site, Kysucké Nové Mesto
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Trnava
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Houghton Gauteng
- Taiwan (3):
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Taipei
- Research Site, Bangkok, Thailand